CLINICAL TRIAL: NCT05291000
Title: The Role of Training And Medication Reminder Wristwatch in the Adherence to The Treatment in Geriatric Patients Diagnosed With Hypertension: A Randomized Controlled Trial (RoT-ReWiH)
Brief Title: The Role of Training and Reminder Wristwatche in Hypertension
Acronym: RoT-ReWiH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Birsen ALTAY, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 83116987-662
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hypertension; Adherence, Medication
Keywords: Elderly; Hypertension; Treatment Adherence; Training; Medication Reminder
MeSH Terms: conditions — Hypertension; Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RoT-ReWiH (Experimental): First, pre-tests were applied to the patients in the training and reminder by watch group at first home visit.Second home visits were conducted participants 12th weeks after the first home visit.One of the researchers presented the education program to individuals with hypertensive.The education program included issues related to hypertension, measurament of pressure blood, lifestyle changes and adherence to treatment. The program using face-to-face communication technique and lasted about 45 minutes.For the patients in this group, the alarm time was set according to the time when blood pressure medication was taken, the cord was adjusted according to the arm, and then information was given about the use of the watch. At the end of the interview, the blood pressure of the experimental groups was measured and the measurement value was recorded on the blood pressure follow-up card.
  Interventions: Behavioral: The Role of Training and Reminder Wristwatche in Hypertension (RoT-ReWiH)
- Training group (Experimental): First, pre-tests were applied to the patients in the training group at first home visit.The education program included issues related to hypertension, measurament of pressure blood, lifestyle changes and adherence to treatment. The program using face-to-face communication technique and lasted about 45 minutes. In addition, other drugs used by individuals at home (such as painkillers, antibiotics) were also evaluated during the home visit, and a red label was made on the antihypertensive drug box to distinguish antihypertensive drugs from other drugs. At the end of the interview, the blood pressure of the experimental groups was measured and the measurement value was recorded on the blood pressure follow-up card.
  Interventions: Behavioral: The Role of Training and Reminder Wristwatche in Hypertension (RoT-ReWiH)
- Control group (No Intervention): Pre-tests was applied to the patients in the control group.No intervention was be applied to the patients in this group and second home visit 12th weeks after the first home visit and were readministered the post-tests.

INTERVENTIONS:
Behavioral: The Role of Training and Reminder Wristwatche in Hypertension (RoT-ReWiH) — The present study revealed that multiple interventions such as home visits to elderly hypertensive patients, training program, telephone counseling, and the use of medication reminder wristwatch are effective in increasing treatment adherence and self-efficacy, and in controlling blood pressure. In this direction, health professionals working in primary care are recommended that they make regular home visits, encourage patients to take responsibility for health, and organize regular and interdisciplinary training and counseling programs in the management of hypertension.
  Arms: RoT-ReWiH; Training group

SUMMARY:
This study is a randomized controlled study. The study was completed to with randomized selected 30 training and reminder by watch (experiment), 30 education (experiment) and 30 control group total of 90 hypertensive patients. Patients in the experimental group received training on hypertension and treatment adherence. In addition, the participants in the training and reminder by watch group wore a medication reminder wristwatch. Statistically significant differences were found in the post-test between scale scores of the experimental and control groups (p<.05). It was observed that the initial blood pressure measurements were high in the patients in all three groups, while the highest decrease was found in the training and reminder by wristwatch group at the final measurement (p<.05). Hypertension education program and using a medication reminder wristwatch were found to be effective in increasing treatment adherence.

DETAILED DESCRIPTION:
Design and Participants This study was conducted a randomized controlled trial. The population of the research was the patients who received service from this center, who were 65 years of age and older, who had hypertension, and who were using at least one antihypertensive drug (n=90). Power analysis was conducted to determine the sample size; it was based on the difference in Compliance with Drug Therapy Scale mean scores of hypertensive patients from previous studies.16 The sample size of at least 60 individuals was calculated by taking α = 0.05, power = 0.99, and effect size = 0.863. Keeping in mind that the number of participants may decrease during the study owing to factors such as a health problems or die , 90 subjects were included in the study.

Participants were randomized to medication reminder wristwatch group (n = 30), training group (n = 30) and control (n = 30) groups. In randomization, participants were stratified participants was ensured through the use of stratified sampling method. The patients in all three groups were stratified according to gender (female, male). The patients who were 65 and older, who were diagnosed with hypertension, who used at least one antihypertensive drug, who are literate and open to communication and cooperation, who had blood pressure of 140/90mmHg or above prior to the research, who had a score of 8 and above from the Compliance with Drug Therapy Scale, and who were willing to participate were included in the study. The patients who met the inclusion criteria constituted the sample of the study.

A questionnaire form, Hypertension Information Form (HIF), Antihypertensive Medication Treatment Adherence Scale (AMTAS), Medication Adherence Self-Efficacy Scale Short Form (MASES-SF) were used to collect data. The questionnaire form was developed by using relevant literature and included 33 closed-ended questions about the sociodemographic, health/disease and treatment compliance characteristics of elderly individuals.

Hypertension Information Form (HIF) was prepared by the researcher in line with the literature in order to measure the effectiveness of the hypertension education program. It contains 26 statements about drug use, blood pressure monitoring, and disease management. The questions are Yes/No questions. The "yes" answers receive 1 point, while the "no" answers receive 0 point. The maximum score that can be obtained from the form is 26. A score of 13 and above indicates that patients' knowledge level about hypertension has increased. The current study found Cronbach α = 0.77.

AMTAS is a questionnaire developed by Morisky et al to evaluate medication adherence of individuals with hypertensive in 2003. The scale includes 9 statements to diagnose the medication behavior and the total score varies between 1 and 13. Individuals with a score between 1 and 7 are defined as compliant with treatment, while individuals with a score of 8 and above are defined as non-compliant with treatment. The Turkish version of the AMTAS was validated by Demirezen et al with Cronbach α = 0.82. In this study, the Cronbach's alpha of the scale was determined as 0.51.

MASES-SF was developed in 2012 by Hacıhasanoğlu et al and include of 13 questions on a Likert scale. The total score of the scale is between 13 and 52, and an increase in the score indicates that the individual's level of compliance with antihypertensive drug treatment is good. The Cronbach's alpha was reported as 0.94. In this study, the Cronbach's alpha of the scale was found to be 0.83.

The study was conducted between April 2019 and November 2020. In the first meeting, The questionnaire form, HIF, AMTAS, MASES-SF were administered. Data were collected using the face-to-face interview method.

Ethical approval was obtained from the ethical board (February 18, 2018, No. 83116987-662) and permission was given from the Provincial Health Directorate (February 28, 2019, No. 87064461-044). Participants were informed about the scope of the study and verbal and written informed consent was obtained. Educational material was given to participants of the control group after the last home visit.

The data were analyzed using the SPSS 23.0. Chi-square and Fisher's Exact Tests were used to compare the categorical variables across the groups. One-way Analysis of Variance was used to compare the data that show normal distribution according to groups of three or more, and the Kruskal Wallis Test was used to compare data that were not normally distributed. The paired two-sample t-test was used to compare normally distributed data according to paired time, and the Wilcoxon Test was used to compare the data that did not show normal distribution. The McNemar Test was used to compare the categorical variables according to pretest and posttest. For statistical significance, P < .05 was used.

ELIGIBILITY:
Inclusion Criteria:

-The patients who were 65 and older, who were diagnosed with hypertension, who used at least one antihypertensive drug, who are literate and open to communication and cooperation, who had blood pressure of 140/90mmHg or above prior to the research, who had a score of 8 and above from the Compliance with Drug Therapy Scale, and who were willing to participate were included in the study.

Exclusion Criteria:

* Being diagnosed with malignancy
* İlliteracy
* Having a history of cardiac intervention in the past year
* Hearing-vision loss

Ages: 65 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Antihypertensive Medication Treatment Adherence Scale (AMTAS) | 3 Month
  AMTAS is a questionnaire developed by Morisky et al to evaluate medication adherence of individuals with hypertensive in 2003. The scale includes 9 statements to diagnose the medication behavior and the total score varies between 1 and 13. Individuals with a score between 1 and 7 are defined as compliant with treatment, while individuals with a score of 8 and above are defined as non-compliant with treatment. The Turkish version of the AMTAS was validated by Demirezen et al. with Cronbach α = 0.82. In this study, the Cronbach's alpha of the scale was determined as 0.51.
Medication Adherence Self-Efficacy Scale Short Form (MASES-SF) | 3 Month
  MASES-SF was developed in 2012 by Hacıhasanoğlu et al and include of 13 questions on a Likert scale. The total score of the scale is between 13 and 52, and an increase in the score indicates that the individual's level of compliance with antihypertensive drug treatment is good. The Cronbach's alpha was reported as 0.94. In this study, the Cronbach's alpha of the scale was found to be 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen ALTAY, Doç. Dr., Study Director — Ondokuz Mayıs University
Locations (1):
- Erbaa Family Health Center, Tokat Province, Erbaa, Turkey (Türkiye)